CLINICAL TRIAL: NCT06371183
Title: A Comparative Study of Clinical, Endoscopic and Histopathological Features of Colitis in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Omar Mahmoud Said, AOMSaid, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOMSaidB
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Role of Ileoscopy in Diagnosis of Colitis
MeSH Terms: interventions — Colonoscopes

STUDY DESIGN:
Intervention Model Description: Patients who complaining of lower GI manifestations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with lower GI manifestations (Other): Patients with lower GI manifestations will undergo total colonoscopy with biopsy
  Interventions: Device: Colonoscope

INTERVENTIONS:
Device: Colonoscope — Endoscopy for lower GIT

SUMMARY:
A Comparative study of clinical, endoscopic and histopathological features of colitis in children

DETAILED DESCRIPTION:
To find out the role of ileoscopy in diagnosis of colitis and compare clinical , endoscopic and histopathological manifestations of colitis

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients diagnosed as colitis during the study period. 2. Age from 1 month to 18 years.

Exclusion Criteria:

1. Patients with lower gastrointestinal manifestations and weren't diagnosed as colitis during colonoscope.
2. Patients less than one month and more than 18 years.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Is ileoscopy indicated for all children complaining of colitis on 196 patient | 2years
  Biopsy from ileum will be taken to diagnose colitis

SECONDARY OUTCOMES:
To correlate clinical manifestations by colonoscopic picture | 2years
  Some patients with lower GI manifestations,their colonoscopy is normal. So corolate clinical with biopsy

IPD SHARING:
Plan to Share IPD: Undecided
I will share the IPD results